CLINICAL TRIAL: NCT01064518
Title: A Phase 2, Double-Blind, Randomized, Parallel-Group, Controlled, Multi-Center Study to Evaluate the Efficacy and Safety of RT001, a Botulinum Toxin Type A Topical Gel, for the Treatment of Moderate to Severe Lateral Canthal Lines in Adults
Brief Title: Efficacy and Safety Study of RT001 for the Treatment of Moderate to Severe Lateral Canthal Lines in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RT001-CL024LCL
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Lateral Canthal Lines; Crow's Feet; Facial Wrinkles
Keywords: Lateral Canthal Lines; Crow's Feet Wrinkles; Facial Wrinkles
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose A (Active Comparator): RT001 Topical Gel
  Interventions: Drug: Botulinum Toxin Type A
- Dose B (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo (Dose B)

INTERVENTIONS:
Drug: Botulinum Toxin Type A — RT001 (Botulinum Toxin Type A Topical Gel, Dose A) applied topically at Baseline (Day 0) to the lateral canthal lines
  Arms: Dose A
Drug: Placebo (Dose B) — Placebo (Dose B), applied topically at Baseline (Day 0) to the lateral canthal lines
  Arms: Dose B

SUMMARY:
The purpose of this study is to find out if an investigational drug, called RT001 Botulinum Toxin Type A Topical Gel, is safe and useful in minimizing the wrinkles between the eye and hairline called crow's feet, also known as lateral canthal lines.

DETAILED DESCRIPTION:
RT001, a new drug, may be effective for the temporary improvement in the appearance of moderate to severe lateral canthal lines (crow's feet wrinkles) in adults. In this study, researchers want to find out if RT001is more effective than placebo gel by examining the effect on the improvement of crow's feet by both the patient and physician.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent including authorization to release health information
* Female or male, 18 to 65 years of age and in good general health
* Willing and able to follow study instructions and likely to complete all study requirements
* Moderate to severe lateral canthal lines (crow's feet wrinkles)

Exclusion Criteria:

* Any neurological condition that may place the subject at increased risk with exposure to Botulinum Toxin Type A, including peripheral motor neuropathic diseases such as amyotrophic lateral sclerosis and motor neuropathy, and neuromuscular junctional disorders such as Lambert-Eaton syndrome and myasthenia gravis
* Muscle weakness or paralysis, particularly in the area receiving study treatment
* Active disease or irritation at the treatment areas including the eye and the skin
* Pregnant, nursing, or planning a pregnancy during the study; or is a woman of childbearing potential (WOCBP) but is not willing to use an effective method of birth control
* Previous participation in a RT001 clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The number of subjects who show improvement based on the investigator global and patient assessments. | Week 4

SECONDARY OUTCOMES:
The number of subjects who show improvement based on the investigator global and patient assessments. | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Fredric Brandt, MD, Principal Investigator — Dermatology Research Institute, LLC
Locations (1):
- Dermatology Research Institute, LLC, Coral Gables, Florida, United States